CLINICAL TRIAL: NCT03204526
Title: Safety and Feasibility of Using Low Frequency Deep Brain Stimulation of the Subthalamic Nucleus to Improve Cognitive Performance in Patients With Parkinson's Disease
Brief Title: Low Frequency Deep Brain Stimulation of the Subthalamic Nucleus in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 693382
Record Dates: First submitted 2016-12-09; First posted 2017-07-02 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease; Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Deep Brain Stimulation

ARMS (1):
- low frequency stimulation (LFS) (Experimental): Low-frequency deep brain stimulation of the subthalamic nucleus
  Interventions: Device: deep brain stimulation

INTERVENTIONS:
Device: deep brain stimulation

SUMMARY:
Prospective trial of low frequency deep brain stimulation of the ventral subthalamic nucleus to improve cognitive performance in patients with advanced Parkinson's disease. All study participants have undergone DBS implantation surgery as part of their routine care for motor manifestations of Parkinson's disease. In this study, a temporary low frequency period of stimulation will be applied to determine its effects on cognition.

DETAILED DESCRIPTION:
In this randomized cross-over pilot study, our primary aim was to determine the effect of theta (5 Hz), and gamma (130 Hz) frequency stimulation in the ventral STN on cognitive control in patients with PD. This study provides a first look at frequency dependent modulation of cognitive function and provides important insights into the utility of DBS for non-motor symptoms of PD and other neuropsychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease, undergoing deep brain stimulation implantation as part of their routine management of motor symptoms.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Frequency Stimulation (LFS): Low-frequency deep brain stimulation of the subthalamic nucleus
  deep brain stimulation
Period: Overall Study
Arm/Group | Low Frequency Stimulation (LFS)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Frequency Stimulation (LFS)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Year] | 62.18 (6.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Disease Duration [Mean (Standard Deviation); unit: Year] | 7.73 (3.38)

OUTCOME MEASURES:

1. Primary Outcome: Mean Reaction Time for Computerized Color Naming Stroop Task
Description: The Stroop Color and Word Test (SCWT) is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect.
Time Frame: 2 days
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Low Frequency Stimulation (LFS)
Number analyzed (Participants) | 15
seconds | 5.09 [2 to 18]

2. Primary Outcome: Mean Accuracy Rates Using Computerized Color Naming Stroop Task
Description: as for outcome 1
Time Frame: 2 days
Measure: Mean (95% Confidence Interval); unit: percent correct response
Arm/Group | Low Frequency Stimulation (LFS)
Number analyzed (Participants) | 15
percent correct response | 4.61 [2 to 20]

3. Secondary Outcome: Number of Participants With Worsening Depression Using Beck's Depression Index
Description: Questionnaire with numerical score indicating level of depression. Individual scale items are scored on a 4-point continuum (0=least, 3=most), with a total summed score range of 0-63. Higher scores indicate greater depressive severity.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Frequency Stimulation (LFS)
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: Number of Participants Showing Motor Worsening Using the Unified Parkinson's Disease Rating Scale (UPDRS-III)
Description: The UPDRS scale is a rating tool used to gauge the course of Parkinson's disease in patients and consists of the following five segments: 1) Mentation, Behavior, and Mood, 2) ADL, 3) Motor sections, 4) Modified Hoehn and Yahr Scale, and 5) Schwab and England ADL scale.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Frequency Stimulation (LFS)
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Time Frame: Study duration (maximum of 2 months)
Description: No Adverse Events
Arm/Group | Low Frequency Stimulation (LFS)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03204526/Prot_SAP_000.pdf
  • Informed Consent Form (2015-05-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT03204526/ICF_001.pdf